CLINICAL TRIAL: NCT04362852
Title: The Manton Center for Orphan Disease Research Gene Discovery Core (GDC)
Brief Title: Patient Forward Access to Clinical and Technological Research: Genetic Influences on Cancer and Atopic Dermatitis
Acronym: PFACTR02
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Pankaj Agrawal, Associate Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: PFACTR02
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Eczema/Atopic Dermatitis; Cancer
Keywords: lung cancer; atopic dermatitis; eczema; genetic testing; genomics; genomic profiling; whole exome; social media; patient centered
MeSH Terms: conditions — Eczema; Dermatitis, Atopic; Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood or saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer: No intervention
- Atopic Dermatitis/Eczema: No intervention

SUMMARY:
This Patient Forward study intends to conduct research to investigate potential genetic factors causing cancer and eczema/atopic dermatitis. The study utilizes a patient-centered design and is led by a collaborative team including The Manton Center for Orphan Disease Research, Inspire, Citizen Genetics and Pfizer. The Manton Center for Orphan Disease Research, a research program at Boston Children's Hospital that focuses on determining the genetic causes of rare and undiagnosed disorders, will work collaboratively with Inspire (inspire.com), a patient-focused research platform and social network with millions of users, to identify and recruit patients and family members for this genetic research study. Participants for this study will be asked to provide health information through surveys, questionnaires and/or interviews, and to provide a genetic sample through a blood draw or saliva sample. The study intends to combine this information to learn more about the genetic drivers in cancer and eczema/atopic dermatitis.

DETAILED DESCRIPTION:
Inspire will survey its members who have eczema/atopic dermatitis or have had cancer to identify patients that match the health criteria for the study including 1) a diagnosis of one of the two diseases under investigation, and 2) evidence of a family history of the disease. Participants will be referred to the Manton Center by Inspire for outreach and consent. After consenting to participation, participants will be asked to participate in the study by providing 1) relevant medical information/records and family history and 2) a blood/saliva/DNA sample for genetic analysis.

The health and family history information allows the investigators to gain a better understanding of the specific disease symptoms seen in an individual or family. The blood/saliva sample is used to obtain DNA which can then be analyzed to identify if there may be a genetic basis of disease pathophysiology using various tools including exome genomic sequencing, genetic variant analysis, familial genotyping and cross-mapping with disease phenotype and severity.

This study will be ongoing for an indefinite period of time, and participation is continuous unless an individual requests to be removed from the study. Participants can request to withdraw at any time. Active participation primarily takes place at the time of enrollment and on a case-by-case basis thereafter for providing clinical updates and/or additional samples. Risks include those associated with routine blood draws/saliva sample collections and emotional distress associated with genetic and/or medical research. Risks are minimized as much as possible by an open consent process and privacy/confidentiality safeguards, including a certificate of confidentiality from the NIH and the use of de-identified, numerical codes to refer to participants with collaborators.

Although there may not be immediate, direct benefits to participants, the possible benefits of this study include: 1) the development of new diagnostic tests and more detailed prognostic information for participants and their families and their disease-linked patient communities and 2) a better understanding of the pathophysiology of these conditions, leading to the development of new potential treatments. Furthermore, this study offers to return genetic test results that are unrelated to cancer and eczema/atopic dermatitis, but are results that may impact health, like an inherited risk for cancer. The American College of Medical Genetics (ACMG) has recommended that findings identified in a subset of medically actionable genes associated with various inherited disorders be reported for those undergoing genomic sequencing. Pathogenic findings in this subset of genes will be returned to the participant.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of eczema or atopic dermatitis and/or being related to a person with such a diagnosis
* Having a past diagnosis of cancer and/or being related to a person with such a diagnosis

Exclusion Criteria:

* Not having such a diagnosis and/or not be related to such an individual

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with eczema/atopic dermatitis or a past cancer diagnosis and their family members
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Identification of novel genetic factors causing cancer or eczema/atopic dermatitis | 1-10 years
  Analysis of genetic data from families impacted by lung cancer or eczema/atopic dermatitis. This may include functional analysis such as animal modeling and cell line assays, which will be performed to gain further insight into novel candidate genes. When a molecular diagnosis is identified for a family, this is reported back through a designated health care provider.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hopsital, Boston, Massachusetts, United States

REFERENCES:
- See also: The Manton Center for Orphan Disease Research — http://www.childrenshospital.org/research/centers-departmental-programs/manton-center-for-orphan-disease-research
- See also: Patient-focused research platform and social network — http://inspire.com